CLINICAL TRIAL: NCT06935890
Title: Jack Jumper Ant Venom Immunotherapy Long-term Effectiveness Investigation
Acronym: JAVELIN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NACE-004
Record Dates: First submitted 2025-04-02; First posted 2025-04-20 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-09

CONDITIONS: Allergy; Immunotherapy; Venom Allergy
Keywords: Jack Jumper Ant; Venom Immunotherapy; Sting challenge; VIT
MeSH Terms: conditions — Hypersensitivity; Venom Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants who have completed Jack Jumper Ant Venom Immmunotherapy treatment (Experimental)
  Interventions: Other: Jack Jumper Ant Venom Immunotherapy

INTERVENTIONS:
Other: Jack Jumper Ant Venom Immunotherapy — Jack Jumper Ant Venom Immunotherapy involves injections, under the skin, of gradually increasing doses of insect venom. The treatment is usually between 3-<6 years duration. Participants will have completed this treatment at least 18 months prior to their enrolment in this trial.

SUMMARY:
Jack Jumper ant (JJA) venom allergy is a uniquely Australian medical condition. It is the leading cause of venom allergy and affects up to three per cent of the population. 70 percent of people with JJA allergy will have another reaction on a repeat sting and this sensitivity appears to persist for many years.

Venom immunotherapy (VIT) has been shown to be a safe and effective treatment in the prevention of severe systemic allergic reactions (anaphylaxis) to future stings. It is currently offered to patients as standard care in Tasmania, South Australia and Victoria. However, whilst JJA VIT has been used for many years, there is a lack of evidence on the long-term benefit of the treatment and how it impacts patient quality of life.

This trial will offer patients who have completed a JJA VIT program (between 3 and < 6-years duration) and have been off-treatment for at least 18-months and < 5 years, to have a supervised JJA sting challenge and blood test to assess their JJA venom tolerance level. It will also ask them to complete a set of questionnaires at different timepoints to obtain a history of their exposure and reactions to JJA stings outside of the hospital setting (field stings), and to measure the impact of the completed VIT and knowledge of their sting challenge outcome on their quality of life and their behaviours around auto-injectors.

These measures will be used to explore the long-term effectiveness of JJA VIT and the impact of a sting challenge post VIT on a patient's quality of life.

DETAILED DESCRIPTION:
This will be a prospective, multicentre, phase 4 clinical trial examining the long-term effectiveness (measured by response to an in-hospital JJA sting challenge, primary outcome) and impact on quality of life of JJA VIT involving 3 Australian tertiary hospital sites offering this treatment - Royal Hobart Hospital, Royal Adelaide Hospital and Monash Medical Centre.

Patients who have completed their JJA VIT (between 3 and <6 years duration) at one of the 3 sites and off-treatment for at least 18 months and < 5 years, will be invited to participate in the trial by their original treating site. A research team member will obtain informed e-consent and a booking for an in-clinic JJA sting challenge will be allocated. For all consented participants, quality of life (QoL), anxiety and depression scores, history of field sting reactions since treatment completion and attitudes toward adrenaline autoinjector carriage/usage will be collected via questionnaire at trial enrolment, sting challenge, 1-month post sting challenge and annually for 3-years. A blood sample will be collected immediately prior to the sting challenge at the in-clinic appointment. Participants will also be asked to consent to access retrospective data related to their completed JJA VIT course from their hospital clinical records.

Optional consents will also be sought from each participant for the collection of an extra tube of blood with the serum biobanked for future analysis, and the inclusion of their data in the National Allergy BioRepository (ALBI).

ELIGIBILITY:
Eligibility criteria

- Any adult (≥ 18 years) who has completed a JJA VIT program at one of the three participating sites.

Inclusion Criteria:

1. Completed a continuous program of JJA VIT of between 3 and < 6 years duration.
2. Have ceased JJA VIT for ≥ 18 months but < 5 years.
3. Have the ability to provide informed consent.

Exclusion Criteria:

1. Any person < 18 years.
2. Any adult (≥ 18 years) who has not completed a continuous JJA VIT program of duration between 3 and < 6 years.
3. Any adult (≥ 18 years) who has completed a continuous JJA VIT program of duration between 3 and < 6 years but ceased JJA VIT < 18 months or > 5 years ago.
4. Any person who has a medical condition, that in the opinion of the investigator, may place them at increased risk if they were to have a sting challenge.
5. Unable to understand study requirements and provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Presence of systemic reaction as assessed by the clinician | Periprocedural
  This will be recorded by the clinician as YES or NO.
Severity of a clinically assessed systemic reaction measured by The Brown Grading Criteria | Periprocedural
  The Brown Grading Criteria measures the severity of anaphylactic reactions by categorizing symptoms based on body systems affected and physiological impact. The tool uses a 3-point grading system: Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe. Higher scores indicate more severe anaphylactic reactions.

SECONDARY OUTCOMES:
Change in presence of a systemic reaction to a field sting following cessation of Jack Jumper Ant Venom Immunotherapy as reported by the patient on a trial-specific questionnaire | At enrolment, 1-month post procedure and annually for 3-years
  Trial specific questionnaire to be completed by the patient which captures information about any Jack Jumper Ant stings that the patient may have had since completion of Venom Immunotherapy Treatment and whether or not they experienced any type of reaction. If no sting was experienced only one question is required to be answered. If sting/s was experienced ten questions are asked including timing, symptoms, location, treatment and environment.
Change in severity of a systemic reaction to a field sting following cessation of Jack Jumper Ant Venom Immunotherapy as measured by The Brown Grading Criteria | At enrolment, 1-month post procedure and annually for 3-years
  The Brown Grading Criteria measures the severity of anaphylactic reactions by categorizing symptoms based on body systems affected and physiological impact. The tool uses a 3-point grading system: Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe. Higher scores indicate more severe anaphylactic reactions.
Change in attitude towards adrenaline auto-injectors as measured by the Adrenaline Auto-injector Questionnaire | At enrolment, 1-month post procedure and annually for 3-years
  The Adrenaline Auto-injector Questionnaire measures patient attitudes and behaviors related to adrenaline auto-injectors as a 4 question survey. Current possession of an adrenaline auto-injector (yes/no), decision-making process regarding auto-injector maintenance (doctor advice, personal decision, or other influence), carrying/storage behaviors (ranging from constant carriage to unknown location), overall attitude assessment using a 7-point scale regarding the advantages and disadvantages of carrying an auto-injector where the minimum score is 1 and the maximum score is 7. A lower score indicates a better outcome.
Change in quality of life as measured by the Vespid Quality of Life Questionnaire | At enrolment, 1-month post procedure and annually for 3-years
  An adapted insect allergy specific health-related quality of life questionnaire.
  14 questions with 7 response options giving a score of 1-7, with lower scores representing a higher quality of life.
Change in quality of life measured using the Hospital Anxiety and Depression Scale | At enrolment, 1-month post procedure and annually for 3-years
  Developed to assess depression and anxiety. Each response ranges from 0 to 3, the 14 responses are added to yield a total score between 0 and 42. Higher scores indicate higher severity of anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Le, MBBS FRACP, Principal Investigator — Royal Hobart Hospital
Locations (3):
- Australia (3):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Medical Centre, Clayton, Victoria

IPD SHARING:
Plan to Share IPD: Yes
After the data has been cleaned and database has been locked, the de-identified data and if consented, personal identifying information, will be shared to National Allergy Centre of Excellence (NACE) Allergy BioRepository via a safe and secure mechanism, for storage and use in future allergy research.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: At 6 months post the commencement of JAVELIN, de-identified data, encrypted with NACE unique identifier codes and secure linkage key tokens, will be transferred to the ALBI platform, for storage, integration and sharing for future HREC-approved allergy research purposes. Data once in ALBI remains indefinitely.
Access Criteria: ALBI will only provide researchers with non-identifiable information following the Scientific Access Framework. Researchers need to apply for access to ALBI data. Once approved, data will be made available to the researchers by logging in through a secure research platform. Researchers will not have access to the entire ALBI system as they will be provided extracts from ALBI of non-identifiable information related to their specific request and approval. Information will only be shared with ethically approved future allergy research studies.
URL: https://www.nace.org.au/

REFERENCES:
- See also: JAVELIN trial information — https://www.nace.org.au/research/insect-allergy/